CLINICAL TRIAL: NCT05391997
Title: Comparative Effects of Cervical Extension Traction Exercises With and Without Modified Cervical and Shoulder Retraction Exercises on Pain, Disability and Cobb's Angle in Patients With Non-specific Neck Pain
Brief Title: Effects of Cervical Extension Traction With & Without Modified Cervical and Shoulder Retraction Exercises in Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0117
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Neck Pain
Keywords: neck pain; retraction; disability; cervical traction
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Cervical and Shoulder Retraction exercises (Experimental): Cervical extension traction protocol will be added as standard treatment. Then, patients either sit or stand in an upright position while pushing their chin backward and simultaneously raising their head within the pain-free range, then, in a seated or standing position, patients will maintain an upright posture and try to pull back their shoulders and extend their neck within the pain-free range.
  Interventions: Other: Modified Cervical and Shoulder Retraction exercises
- Cervical Extension Traction exercises (Active Comparator): Here, patients will receive Cervical Extension Traction exercises as standard treatment. Cervical extension traction includes a protocol in which traction will be applied within the extension range of the cervical region in full spine position.
  Interventions: Other: Cervical Extension Traction exercises

INTERVENTIONS:
Other: Modified Cervical and Shoulder Retraction exercises — 11 patients will receive cervical traction and modified cervical and shoulder retraction exercises (10 to 12 repetitions). The total treatment session will be of 20-25 minutes with a total intervention period of 6 weeks with 3 sessions per week on alternative days.
  Arms: Modified Cervical and Shoulder Retraction exercises
Other: Cervical Extension Traction exercises — 11 patients will receive cervical traction force for 10 seconds and extend the cervical spine. The total treatment session will be of 20-25 minutes with a total intervention period of 6 weeks with 3 sessions per week on alternative days
  Arms: Cervical Extension Traction exercises

SUMMARY:
The study aims to explore whether the modified cervical and shoulder retraction exercise program restores cervical sagittal alignment and reduces neck pain in patients with non-specific neck pain.

DETAILED DESCRIPTION:
Neck pain is a musculoskeletal system disorder that causes social and economic loss by reducing the quality of life (QOL) of the individual, and its prevalence varies from 16.7 to 75.1% in the adult population. Non-specific neck pain (NNP) is a symptom related to a postural or mechanical cause. NNP is also associated with loss of cervical curvature. In healthy spines, the axial load along the cervical spine is supported along the ventral column of the spine. However, in spines with the loss of lordosis, the load moves more anteriorly, which causes neck pain. Cervical exercise has been shown to be an effective treatment for neck pain and cervical alignment, but there is still a need for more clinical trials evaluating the effectiveness of the exercise approach. It seems reasonable to assume that naturally good neck muscle strength and range of motion are likely to be protective factors against neck pain.

As per previous research, the effects of exercise therapy on non-specific neck pain have been examined but there is limited literature available for use of cervical and shoulder retraction exercises in patients with nonspecific neck pain. Most of the studies have been done with neck isometrics, manual mobilization, and deep cervical flexors training and there is less scope of practicing cervical extension traction in contrast with modified cervical and shoulder retraction exercises. Previous research is limited by no use of a control group in a modified retraction exercise regime. To fill this literature gap this study is proposed which will focus on the clinical significance of modified cervical and shoulder retraction exercises on pain, disability, and Cobb's angle in the management of non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain history
* Patients with Lateral Cervical Radiograph
* Patients who agreed for a follow up of 6 weeks

Exclusion Criteria:

* Congenital abnormalities e.g. torticollis
* Past surgical history of cervical spine
* Positive VBI sign
* Patients with inflammatory or rheumatic diseases
* Already undergoing physiotherapy treatment

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 6th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
NDI for disability | 6th week
  The neck disability index (NDI) has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. The maximum score is 50
Lateral cervical radiograph for Cobb's angle | 6th week
  Radiography of a patient provides important spine/posture data, such as segmental and total angles of curvature and sagittal balance. Cobb's angle measurement taken by Lateral Cervical Radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Physiotherapy department Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sbardella S, La Russa C, Bernetti A, Mangone M, Guarnera A, Pezzi L, Paoloni M, Agostini F, Santilli V, Saggini R, Paolucci T. Muscle Energy Technique in the Rehabilitative Treatment for Acute and Chronic Non-Specific Neck Pain: A Systematic Review. Healthcare (Basel). 2021 Jun 17;9(6):746. doi: 10.3390/healthcare9060746. PMID 34204590
- [Background] Paolucci T, Agostini F, Mangone M, Bernetti A, Cordiani B, Bellomo RG, Saggini R, Villani C. Sagittal spine alignment and postural balance in pre-puberty age: a multidisciplinary and multi-professional rehabilitative point of view. J Biol Regul Homeost Agents. 2021 Jan-Feb;35(1):367-372. doi: 10.23812/20-621-L. No abstract available. PMID 33511839
- [Background] Lee MY, Jeon H, Choi JS, Park Y, Ryu JS. Efficacy of Modified Cervical and Shoulder Retraction Exercise in Patients With Loss of Cervical Lordosis and Neck Pain. Ann Rehabil Med. 2020 Jun;44(3):210-217. doi: 10.5535/arm.19117. Epub 2020 May 29. PMID 32475094
- [Background] de Zoete RM, Armfield NR, McAuley JH, Chen K, Sterling M. Comparative effectiveness of physical exercise interventions for chronic non-specific neck pain: a systematic review with network meta-analysis of 40 randomised controlled trials. Br J Sports Med. 2020 Nov 2:bjsports-2020-102664. doi: 10.1136/bjsports-2020-102664. Online ahead of print. PMID 33139256
- [Background] Multanen J, Hakkinen A, Kautiainen H, Ylinen J. Associations of neck muscle strength and cervical spine mobility with future neck pain and disability: a prospective 16-year study. BMC Musculoskelet Disord. 2021 Oct 29;22(1):911. doi: 10.1186/s12891-021-04807-3. PMID 34715847
- [Background] Jahre H, Grotle M, Smedbraten K, Dunn KM, Oiestad BE. Risk factors for non-specific neck pain in young adults. A systematic review. BMC Musculoskelet Disord. 2020 Jun 9;21(1):366. doi: 10.1186/s12891-020-03379-y. PMID 32517732
- [Background] Jun D, Johnston V, McPhail SM, O'Leary S. A Longitudinal Evaluation of Risk Factors and Interactions for the Development of Nonspecific Neck Pain in Office Workers in Two Cultures. Hum Factors. 2021 Jun;63(4):663-683. doi: 10.1177/0018720820904231. Epub 2020 Mar 2. PMID 32119582
- [Background] Moustafa IM, Diab AA, Hegazy F, Harrison DE. Demonstration of central conduction time and neuroplastic changes after cervical lordosis rehabilitation in asymptomatic subjects: a randomized, placebo-controlled trial. Sci Rep. 2021 Jul 28;11(1):15379. doi: 10.1038/s41598-021-94548-z. PMID 34321539
- [Background] Oakley PA, Ehsani NN, Moustafa IM, Harrison DE. Restoring cervical lordosis by cervical extension traction methods in the treatment of cervical spine disorders: a systematic review of controlled trials. J Phys Ther Sci. 2021 Oct;33(10):784-794. doi: 10.1589/jpts.33.784. Epub 2021 Oct 13. PMID 34658525
- [Background] Moon H, Lee SK, Kim WM, Seo YG. Effects of exercise on cervical muscle strength and cross-sectional area in patients with thoracic hyperkyphosis and chronic cervical pain. Sci Rep. 2021 Feb 15;11(1):3827. doi: 10.1038/s41598-021-83344-4. PMID 33589667
- [Background] Villanueva-Ruiz I, Falla D, Lascurain-Aguirrebena I. Effectiveness of Specific Neck Exercise for Nonspecific Neck Pain; Usefulness of Strategies for Patient Selection and Tailored Exercise-A Systematic Review With Meta-Analysis. Phys Ther. 2022 Feb 1;102(2):pzab259. doi: 10.1093/ptj/pzab259. PMID 34935963
- [Background] Kashfi P, Karimi N, Peolsson A, Rahnama L. The effects of deep neck muscle-specific training versus general exercises on deep neck muscle thickness, pain and disability in patients with chronic non-specific neck pain: protocol for a randomized clinical trial (RCT). BMC Musculoskelet Disord. 2019 Nov 14;20(1):540. doi: 10.1186/s12891-019-2880-x. PMID 31727085